CLINICAL TRIAL: NCT02656316
Title: The Effects of Multi-focal Transcranial Direct Current Stimulation (tDCS) on Motor-cognitive Dysfunctions and Freezing of Gait in Patients With Parkinson's Disease: A Randomized Controlled Trial
Brief Title: The Effects of Multi-focal tDCS on Motor-cognitive Dysfunctions in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Director of Research and Developmen, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TASMC-15-NIR-710-CTIL
Record Dates: First submitted 2016-01-13; First posted 2016-01-14 (Estimated); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active tDCS (Experimental): The active tDCS condition will consist of 20 min of continuous stimulation. This amount of stimulation is safe for healthy young and older adults and has been shown to induce acute beneficial changes in cortical excitability and cognitive functions.
  Interventions: Device: Active tDCS
- Sham tDCS (Sham Comparator): The Sham tDCS - an inactive stimulation.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — In this group subjects will receive 20 min of treatment.
  Arms: Active tDCS
Device: Sham tDCS — In this group subjects will receive 20 min of sham stimulation.
  Arms: Sham tDCS

SUMMARY:
The current RCT aims to establish the therapeutic potential of tDCS for freezing of gait (FOG) and motor-cognitive dysfunctions in PD. As noted, FOG is often unresponsive to pharmacological and other treatments, especially in the advanced stages of the disease. While it is likely that tDCS will provide symptomatic relief, we will also explore, via secondary outcomes, the potential for tDCS to modify disease progression. Support for this possibility stems from the likely mechanisms of action of tDCS.

DETAILED DESCRIPTION:
The current study aim to establish the therapeutic potential of tDCS for freezing of gait (FOG) and motor-cognitive dysfunctions in Parkinson's Disease (PD). FOG phenomenon is often unresponsive to pharmacological and other treatments, especially in the advanced stages of the disease. While it is likely that Transcranial direct current stimulation (tDCS) will provide symptomatic relief, we will also explore, via secondary outcomes, the potential for tDCS to modify disease progression. Support for this possibility stems from the likely mechanisms of action of tDCS.

Based on strong rationale and preliminary findings in previous works, the objectives of the current proposal are to conduct a prospective multi-center, double-blinded, stratified controlled randomized clinical trial, comparing real multifocal tDCS to sham stimulation. The main aim:

- To demonstrate the "short-term" and the longer-term effects of tDCS on FOG severity and frequency.

Participants: A total of 85 patients will be recruited (Hoehn and Yahr Stage 1-3.5) who suffer from FOG, as measured by the new FOG questionnaire (NFOG-Q) and as demonstrated in response to a FOG provoking protocol, who are on stable medications, who have no contraindications to tDCS, and who are between the ages of 40-80. Patients with DBS will not be included.

tDCS intervention: Subjects will be randomized to receive either a real or sham tDCS intervention. Each intervention will consist of 10, 20-minute treatments completed over 2 consecutive weeks (i.e., 5 per week), following previously established protocols. A single, weekly "maintenance" treatment will then be provided for the following 12 weeks (note: for depression, maintenance tDCS is most often provided once every two weeks; we will take a more conservative approach here in this first long-term study for FOG in PD).

Participants will continue taking their regular medications, and treatments will take place in the "ON" medication state (approximately at the same time of day for each treatment). The real tDCS intervention will simultaneously target both the M1 leg area and the the dorsolateral prefrontal cortex (DLPFC), in the brain hemisphere contralateral to the more affected side of the body, as determined by the summation of the motor symptoms on The unified Parkinson's disease rating scale (UPDRS). Current will be applied using an array of 8 sponge electrodes and the StarStim tDCS device and software (Neuroelectrics, Inc). For this protocol, the placement and current delivered through each electrode has been optimized using the Neuroelectrics StimWeaver® Stimulation Optimization Service . In case of bilateral symptom symmetry, tDCS will target the left M1 and DLPFC. For the sham intervention, the same electrode placement and stimulation parameters will be used; however, current will only be applied for the first 60 seconds of the stimulation session. This is a reliable control as sensations arising from tDCS diminish considerably after the first minute of stimulation. At the end of each treatment session, participants will complete a short questionnaire to assess potential side-effects. At the end of the entire intervention, participants will be asked to state if, in their opinion, they received the real or sham intervention.

Outcome measures: The primary outcome will be the number of FOG episodes measured in the lab when subjects undergo a validated FOG-invoking protocol, after the initial 2-week intervention and at the final study point, similar to that proposed by Ziegler et al. Briefly, this protocol includes situations that have been shown to provoke FOG. Patients will be asked to sit, to stand up and to walk to a a mark on the floor. They will perform two 360° turns, clockwise and counter-clockwise. Then, the patients will be asked to open a door and walk through it, turn outside, and come back to their chair. Secondary outcomes of FOG will include FOG duration and the new FOG questionnaire (NFOG-Q). This FOG-provoking protocol will take place in both the ON and OFF medication state and higher values (worse) of FOG will be used as the primary outcome measure (in secondary analyses, we will examine ON and OFF FOG separately).

Additional secondary measures will test the influence of tDCS on other motor, cognitive or motor-cognitive functions related to PD and FOG. Secondary outcomes related to motor function, which are likely to be affected by changes in M1 excitability, will include gait speed (usual walking), Timed Up & Go scores, UPDRS motor scores, and level of activity over 7 days using portable, lightweight, water-proof sensors. Secondary measures of executive function, which are hypothesized to be responsive to tDCS of the DLPFC, will include the Trail Making test (TMT) parts A and B, and a previously validated computerized neuropsychological battery that provides normalized scores for executive function and attention (and memory). Dual-tasking gait speed (i.e., walking while performing a serial subtraction test) will assess motor-cognitive interactions. Functional near infra-red spectroscopy (available in Boston and Tel Aviv) will assess frontal activation during dual-tasking walking; this reflects the subjects ability to handle cognitive loading and has been associated with FOG. Finally, the PDQ-39 will evaluate quality of life.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria: patients diagnosed with PD, with Hoehn and Yahr Stage between 1-3.5, who suffer from FOG, as measured at screening by the previously validated new FOG questionnaire (NFOG-Q), whose medications have not changed within 1 month of the study and are not anticipated to change during the study, are able to walk independently, and who are between the ages of 40-80 inclusive.

Exclusion Criteria:

Subjects who show no FOG during testing in the lab in response to a FOG provoking protocol, any diagnosed psychiatric or other neurological disorder, stroke, unbalanced and high blood pressure, pregnancy, participation in any clinical trial in the last three months, unwillingness to be randomized; implanted with deep brain stimulation, pacemakers, intracranial electrodes, implanted defibrillators or any other prosthesis; or a perceived inability to complete the study. Additional exclusion criteria related to tDCS safety will include a personal or family history of epilepsy, the use of neuro-active drugs, or risk of metal fragments in the eyes or head.

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Changes in frequency and severity of the freezing of gait phenomenon | short (two weeks) after treatment and long term following (11 weeks) after treatment
  Clinical assessment of freezing of gait: Gait tasks to provoke FOG (e.g. gait trajectory with dual tasking).

SECONDARY OUTCOMES:
Changes in cognitive performance | short (two weeks) after treatment and long term following (11 weeks) after treatment
  The NeuroTrax software uses tests of cognitive performance that measure similar cognitive functions to traditional paper-based tests.
Immediate change in gait mesurments | short (two weeks) after treatment and long term following (11 weeks) after treatment
  Gait speed and variability will be assessed under usual and dual task conditions and while negotiating physical obstacles, using a sensorized 7 meter carpet (PKMAS) and wearable body fixed sensors. These measures will be compared to baseline performance.

CONTACTS AND LOCATIONS:
Overall Officials: Nir Giladi, M.D, Principal Investigator — Head of Neurological institute, Tel-Aviv Sourasky medical center
Locations (1):
- Institute for Aging Research, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Weiss A, Herman T, Giladi N, Hausdorff JM. New evidence for gait abnormalities among Parkinson's disease patients who suffer from freezing of gait: insights using a body-fixed sensor worn for 3 days. J Neural Transm (Vienna). 2015 Mar;122(3):403-10. doi: 10.1007/s00702-014-1279-y. Epub 2014 Jul 29. PMID 25069586
- [Result] Leite J, Goncalves OF, Carvalho S. Facilitative effects of bi-hemispheric tDCS in cognitive deficits of Parkinson disease patients. Med Hypotheses. 2014 Feb;82(2):138-40. doi: 10.1016/j.mehy.2013.11.021. Epub 2013 Dec 1. PMID 24332532
- [Result] Zhou J, Hao Y, Wang Y, Jor'dan A, Pascual-Leone A, Zhang J, Fang J, Manor B. Transcranial direct current stimulation reduces the cost of performing a cognitive task on gait and postural control. Eur J Neurosci. 2014 Apr;39(8):1343-8. doi: 10.1111/ejn.12492. Epub 2014 Jan 20. PMID 24443958
- [Derived] Manor B, Dagan M, Herman T, Gouskova NA, Vanderhorst VG, Giladi N, Travison TG, Pascual-Leone A, Lipsitz LA, Hausdorff JM. Multitarget Transcranial Electrical Stimulation for Freezing of Gait: A Randomized Controlled Trial. Mov Disord. 2021 Nov;36(11):2693-2698. doi: 10.1002/mds.28759. Epub 2021 Aug 18. PMID 34406695